CLINICAL TRIAL: NCT04035538
Title: A Randomized, Open-label, Single-dose, Replicate-crossover Study to Compare the Safety and Pharmacokinetics of CKD-320 and D012 in Healthy Subjects
Brief Title: A Clinical Study to Compare the Safety and Pharmacokinetics of CKD-320 and D012
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A94_01BE1909
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Hypertension
Keywords: CKD-320
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental)
  Interventions: Drug: CKD-320, D012
- B group (Experimental)
  Interventions: Drug: CKD-320, D012

INTERVENTIONS:
Drug: CKD-320, D012 — R: D012 1tablet, QD, PO T: CKD-320 2tablets, QD, PO

SUMMARY:
A clinical study to compare the safety and pharmacokinetics of CKD-320 and D012

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, replicate-crossover study to compare the safety and pharmacokinetics of CKD-320 and D012 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult older than 19 years at the time of screening
2. Body weight more than 55kg and within ±20% of the calculated ideal body weight(IBW = (height -100) x 0.9)
3. No congenital or chronic disease and no pathological symptoms or findings
4. Suitable subject who is determined to be suitable in laboratory testing such as hematology, blood chemistry, urinalysis and 12-lead electrocardiogram
5. Subject who have received a detailed explanation of this clinical trial and have fully understood it, and agree in writing to comply

Exclusion Criteria:

1. Subject who has a history of clinical significant hepatobiliary, kidney, digestive, respiratory, blood-oncology, endocrine, urinary, psychiatric, musculoskeletal, immune, acute and unstable heart failure or evidence
2. Subject with a history of gastrointestinal disorders(Crohn's disease, ulcer, acute or chronic pancreatitis) or gastrointestinal surgery(except for simple appendicitis surgery or hernia surgery) that may affect the absorption
3. A hereditary angioedema patient, with a history angioedema, or hereditary fructose patient
4. Clinical laboratory test results showing the following values

   * ALT or AST > 2 times upper limit of normal range
   * eGFR < 60mL/min/1.73m2
5. Subject with a history of overreaction or clinical significant hypersensitivity to drugs
6. Subject who has a systolic blood pressure > 140mmHg or < 100mmHg, diastolic blood pressure > 90mmHg or < 60mmHg, pulses ≥ 100 per minutes
7. In case of past history of drug abuse or positive for urine test of drug abuse
8. Those taking medication known to significantly induce or inhibit drug metabolizing enzymes within 30days before the first administration of clinical trial drug
9. Those taking prescription drugs, natural drug(ex, St. John's wort), herbal medicine within 14days and non-prescription drugs or vitamin supplements within 7days before the first administration of clinical trial drug
10. Those taking other clinical trial drugs or bioequivalence test drugs within 6months before the first administration of clinical trial drug
11. Those who donated whole blood within 2 months or those who donated the components within 1 month or blood transfusion within 1 month before the first administration of the clinical trial drug
12. Subject who has a history of regular alcohol consumption exceeding 210g/week within 6months of screening (1 glass of beer(5%)=10g, 1 glass of soju(20%)=8g, 1 glass of wine(12%)=12g)
13. > 10 smokers per day within 3months of screening and those who can't quit smoking
14. Blood test(RPR Ab, HBS Ag, HCV Ab, anti HIV(AIDS)) results indicate a positive
15. Subject who can't comply with the lifestyle guidelines
16. A pregnant(a likely), breastfeeding women
17. Subject who don't agree or can't comply reliable contraception from screening to 14days after the last drug administration
18. Subject who is judged by the investigator principal to be ineligible to participate in the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
AUCt of CKD-320 | predose(0 hour), 0.17, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours
Cmax of CKD-320 | predose(0 hour), 0.17, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours

SECONDARY OUTCOMES:
Tmax of CKD-320 | predose(0 hour), 0.17, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours
t1/2 of CKD-320 | predose(0 hour), 0.17, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours
AUCinf of CKD-320 | predose(0 hour), 0.17, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours
AUCt/AUCinf of CKD-320 | predose(0 hour), 0.17, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours

IPD SHARING:
Plan to Share IPD: Undecided